CLINICAL TRIAL: NCT04887051
Title: The Effects of Respiratory-based Telerehabilitation on Physical Performance and Factors Affecting Compliance in Patients With Multiple Sclerosis
Brief Title: The Effects of Respiratory-based Telerehabilitaion in Patients With MS
Acronym: MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Anıl Tosun (Other)
Collaborators: Trakya University (Other)
Responsible Party: Sponsor-Investigator, Dr. Anıl Tosun, Assistant professor, Fenerbahce University
Organization: Fenerbahce University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fenerbahçe Üniversitesi
Record Dates: First submitted 2021-04-18; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis; Telerehabilitation; Compliance, Patient
Keywords: Telerehabilitation, Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Patient Compliance | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- telerehabilitation (Experimental): pre-post telerehabilltation
  Interventions: Other: pulmonory based home exercises

INTERVENTIONS:
Other: pulmonory based home exercises — web based telerehablitation
  Other Names: telerehabilitation

SUMMARY:
During the pandemic, it is important for people who are isolated in their homes to stay inactive and exercise exercises in order to prevent their complaints from increasing due to inactivity. Individuals with multiple sclerosis are outpatient or inpatient with home exercise programs besides the rehabilitation practices. They are being monitored. It has been reported the rehabilitation of individuals is that they need to comply with their home exercise programs in order to contribute. However, very limited research studies suggest that any method can be used as home exercise has examined whether it has increased compliance with the program. However, examining the factors affecting the compliance of individuals with Multiple sclerosis to the home exercise program. The study was not found either.

Exercise through tele-rehabilitation in individuals with multiple sclerosis in previous studies where their education contributed to the physical performance of patients shown. However, these studies are based on individual neurorehabilitation models. In the literature, the use of video-based exercise training in MS patients a study showing increased performance as well as increased participation in the home program available. However, in this study, a special program was applied to the individual and it is not a respiration-based program. There is no research on web-based group activity training in the field.

DETAILED DESCRIPTION:
Multiple sclerosis is chronic and improves the quality of life of the person is a neurological disease that decreases. Multiple Sclerosis in mobility and functional activities cause restrictions in social and professional life, leading to different degrees of disability. It is a disease that causes severe disability and impairs the quality of life. MS, It is one of the most common diseases that cause disability, usually between the ages of 15-50. In recent years, combating disability caused by MS is the most important and has been the main focus. Patients' life expectancy is gradually increasing, One of the important reasons for this is symptomatic treatments and modern rehabilitation. It is said to have applications.

Depression affects approximately 50% of patients with MS. The social isolation caused by quarantine may have increased depression. In MS, in combating spasticity, as well as depression and chronic fatigue, regular exercise is important.

During the pandemic, it is important for people who are isolated in their homes to stay inactive and exercise exercises in order to prevent their complaints from increasing due to inactivity. Individuals with multiple sclerosis are outpatient or inpatient with home exercise programs besides the rehabilitation practices. They are being monitored. It has been reported the rehabilitation of individuals is that they need to comply with their home exercise programs in order to contribute. However, very limited research studies suggest that any method can be used as home exercise has examined whether it has increased compliance with the program. However, examining the factors affecting the compliance of individuals with Multiple sclerosis to the home exercise program. The study was not found either.

Exercise through tele-rehabilitation in individuals with multiple sclerosis in previous studies where their education contributed to the physical performance of patients shown. However, these studies are based on individual neurorehabilitation models. In the literature, the use of video-based exercise training in MS patients a study showing increased performance as well as increased participation in the home program available. However, in this study, a special program was applied to the individual and it is not a respiration-based program. There is no research on web-based group activity training in the field.

ELIGIBILITY:
Inclusion Criteria: ambulatuar or non -ambulatuar

* All patients with diagnosed with Multiple Sclerosis. (Diagnosis of MS according to the revised McDonald Criteria 2017)
* An ability to understand and execute simple instructions.
* Aged 20-65 years old.

Exclusion Criteria:

* patients with hearing, vision and cognitive problems.
* Pregnancy (self-reported)
* Orthopedic and other neurological disorders affecting upper limb movements (e.g., epileptic seizures)
* Contra-indication to physical activity (e.g., heart failure, severe osteoporosis) MS clinical relapse or treatment with corticosteroid therapy within 30 days prior to enrollment
* Started or stopped a disease-modifying therapy for MS within 30 days prior to enrollment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Barthell Scale | 1st assesment: At first day (baseline avaluation); 2nd assesment: Change from baseline BI score at 1 month after the program start. 3rd assesment: Change from baseline BI score at 2 month after the program start
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. Time to administer- Self report: 2-5 minutes; Direct observation: 20 minutes. Each item is rated in terms of whether the patient can perform the task independently, with some assistance, or is dependent on help based on observation (0=unable, 1=needs help, 2=independent). The final score is x 5 to get a number on a 100 point score. Barthel scores are that scores of 0-20 indicate "total" dependency and 91-99 indicates "slight" dependency.
Functional Ambulatation Categories | 1st assesment: At first day (baseline avaluation); 2nd assesment: Change from baseline FAC score at 1 month after the program start. 3rd assesment: Change from baseline FAC score at 2 month after the program start.
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. Functional Ambulation Classification (FAS): FAS is a valid and reliable scale that evaluates the physical support needed during walking over 6 scores between 0 and 5. It is scored according to the support needed by the patient through observation. Accordingly, the scores; 0- It cannot be ambulatory alone, except for the parallel bar, the patient needs the help of at least 2 people in order to be ambulatory. 5- It walks independently on all floors.
Fatigue Severity Scale | 1st assesment: At first day (baseline avaluation); 2nd assesment: Change from baseline FSS score at 1 month after the program start. 3rd assesment: Change from baseline FSS score at 2 month after the program start
  The Fatigue Severity Scale (FSS) is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. Essentially, the FSS consists of answering a short questionaire that requires the subject to rate his or her own level of fatigue. The obvious problem with this measure is its subjectivity.A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. It is simple to understand and takes an average of eight minutes to answer.

CONTACTS AND LOCATIONS:
Overall Officials: Anıl Tosun, Dr., Study Chair — Fenerbahce University; Hilal Keklicek, Asc.Prof., Study Director — Trakya University
Locations (1):
- Fenerbahce University, Istanbul, Turkey (Türkiye)